CLINICAL TRIAL: NCT03452280
Title: Validation of the JADE wRAP™, a Novel Blood Pressure Measurement Device, Using the Same Arm Sequential Method
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Jade Healthcare Group Inc. (Industry)
Collaborators: Allphase Clinical Research Inc. (Unknown)
Responsible Party: Sponsor
Other Study IDs: BP1
Record Dates: First submitted 2018-02-26; First posted 2018-03-02 (Actual); Last update posted 2021-02-11 (Actual); Status verified 2021-02

CONDITIONS: Blood Pressure

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The JADE wRAP™, a wrist worn cuff to measure blood pressure and its supporting software platform is currently at the final alpha prototype stage of development and is not intended for sale.

There are minimal risks with using the JADE wRAP™ device; however, the likelihood of these risks has been reduced through design limitations on electrical power delivered to the device and of the pressure delivered to the cuff portion. Patients should experience little to no discomfort from the inflation of the JADE wRAP™ cuff.

DETAILED DESCRIPTION:
The purpose of this study is to validate the JADE wRAP™ in adult patients (≥18 years of age) according to American National Standard, ANSI/AAMI/ISO 81060-2:2013, Non-invasive sphygmomanometers - Part 2: Clinical investigation of automated measurement type.

The study is intended to be a simple validation of blood pressure parameters only (Systolic and Diastolic). This study is not intended to yield any other special information.

OBJECTIVES

1) To validate the JADE wRAP™ for systolic and diastolic blood pressures compared to the reference standard mercury sphygmomanometer.

The data collected from this study is for internal purposes only and should assist in further developing the device and supporting platform to a beta stage.

ELIGIBILITY:
Inclusion Criteria:

1. Must be at least 18 years of age
2. Male or Female
3. Must provide written informed consent prior to the performance of any study-related procedures.

Exclusion Criteria:

1. Subjects who in the opinion of the study staff are too agitated, distressed or who are otherwise unable to cooperate with study procedures
2. Subjects with bigeminy, trigeminy, isolated ventricular premature beat (VPD) or atrial fibrillation or any other condition, in the opinion of the study staff that can result in a significantly irregular heath rhythm.
3. Subjects with signs or recent history of inflammation or infection of the wrists or at the reference clinical test site.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Gender Distribution
  * 30% Male
  * 30% Female
Study Population: This is a single-center validation study using an auscultatory reference sphygmomanometer (i.e. mercury sphygmomanometer), and shall consist of a minimum of 85 subjects.
Sampling Method: Probability Sample
Enrollment: 140 (Estimated)
Dates: Start 2017-12-18 (Actual); Primary Completion 2021-12-31 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
Validation Criteria 1 | April 30, 2018
  For systolic and diastolic blood pressures, the mean value of the differences of the determinations, of the n individual paired determinations of the JADE wRAPTM and of the observers' determinations with the reference sphygmomanometer for all subjects shall be within or equal to ± 5.0 mmHg (± 0.67 kPa), with a standard deviation, sn, no greater than 8.0 mmHg (1.07 kPa)

SECONDARY OUTCOMES:
Validation Criteria 2 | April 30, 2018
  For the systolic and diastolic blood pressures for each of the m subjects, the standard deviation, sm, of the averaged paired determinations per subject of the JADE wRAPTM and of the observers' determinations with the reference sphygmomanometer shall meet the criteria listed.

CONTACTS AND LOCATIONS:
Overall Officials: Jeff Smith, Principal Investigator — Alio Health Services Inc.
Locations (1):
- Alio Health Services Inc., Ottawa, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No